CLINICAL TRIAL: NCT04284865
Title: Optimizing Maintenance for Patients with Chronic Obstructive Pulmonary Disease Following Pulmonary Rehabilitation Via a Web Platform - Case Study
Brief Title: Optimizing Maintenance for Patients with COPD Via a Web Platform - Case Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Nicole Marquis, adjunct professor, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-3607
Record Dates: First submitted 2020-02-20; First posted 2020-02-26 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2022-06

CONDITIONS: COPD
Keywords: Self-management; Long-term care; Telehealth
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): The web platform includes three respiratory exercises: diaphragmatic breathing, thoracic expansion exercise and thoracic expansion exercise assisted upper limbs. It is suggested to do each of the three exercises once a day (AM and PM), four repetitions each. An electronic logbook is also available on the platform to record the duration and the type of others cardiorespiratory exercise of their choice (cycling, walking, using stairs, etc.) as well as strengthening (upper and lower body).
  Interventions: Other: Web Platform

INTERVENTIONS:
Other: Web Platform — The intervention involves the use of the web platform for 12 months combined with a monthly phone follow-up.

SUMMARY:
Pulmonary rehabilitation (PR) has been shown to improve quality of life of people with COPD by decreasing their symptoms. However, the benefits obtained during PR tend to decrease within six months to one year after PR. The objective of this study is to implement a web platform following PR programs in order to improve COPD patients' adherence to self-management techniques. Therefore, the investigators want to verify whether the addition of a tele-management tool allows the gains obtained during PR to be retained over 3, 6 and 12 months. The hypothesis is that participants will maintain their PR gains if they use the platform.

DETAILED DESCRIPTION:
Introduction: By 2020, chronic obstructive pulmonary disease (COPD) is projected to become the 3rd leading cause of death in the world. Pulmonary rehabilitation (PR) has been shown to improve quality of life of people with COPD by decreasing their symptoms. However, the benefits obtained during PR tend to decrease within six months to one year after PR.

The objective of this study is to implement a web platform following PR programs in order to improve COPD patients' adherence to self-management techniques. Specifically, the investigators will 1) evaluate the adherence to the use of the web platform and 2) the effects on exercise capacity, quality of life, the number of hospitalizations and exacerbations. Therefore, the investigators want to verify whether the addition of a tele-management tool allows the gains obtained during PR to be retained over 3, 6 and 12 months. The hypothesis is that patients will maintain their PR gains if they use the platform.

Methods: Participants with COPD will be selected in a PR group at CHUS Hôtel-Dieu de Sherbrooke. Their initial 10-week rehabilitation program will be followed by the use of a web-based tele-management platform for 12 months. Data will be collected at the beginning of PR (T1), end of the PR (T2), after three months of using the web platform (T3), after six months (Q4) and after 12 months (T5). To measure adherence, the research team will have access to a) the number of connections made on the site, b) the number of exercises performed, c) the duration and type of cardiorespiratory exercises as well as the muscular exercises filled in the logbook and d) the number of exercises performed (breathing, cardiorespiratory and muscular exercises) self-reported by the participants at the time of assessment. For the second objective, the measures used will be FEV1 for lung function, the 6-minutes walk test for exercise capacity, COPD Assessment Test for quality of life, modified BORG scale (0-10) and the medical research center (MRC) for the feeling of dyspnea, the number of hospitalizations over 3, 6 and 12 months (self-reported) and the number of exacerbations via medication taken from their pharmacist.

ELIGIBILITY:
Inclusion Criteria:

* Complete the PR program at CIUSSSS of Estrie-CHUS in Sherbrooke and finishing after December 2019
* To have a mild to very severe diagnosis of COPD (mild: forced expiratory volume in 1 second (FEV1) ) ≥ 80%, very severe: FEV1 <30% and Tiffeneau score <0.7)
* Have a score ≥2 on the Medical Research Council (MRC) dyspnea scale
* Have access to a computer, laptop or cell phone at home with an high speed internet service.

Exclusion Criteria:

* Inability to give informed consent
* Instable condition in the 4 weeks prior to the study (change in medication and symptoms such as dyspnea and sputum (colour and quantity)).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Adherence of each participant | 3 months, 6 months and 12 months
  The number of connections made on the site
Change in Adherence of each participant | 3 months, 6 months and 12 months
  the number of exercises performed on the platform web
Change in Adherence of each participant | 3 months, 6 months and 12 months
  Number of entry/week in the logbook on the platform web
Change in Adherence of each participant | 3 months, 6 months and 12 months
  the number of exercises performed (breathing, cardiorespiratory and muscular exercises) self-reported by the participants

SECONDARY OUTCOMES:
Change in Exercise capacity | pre-pulmonary rehabilitation, 0 months, 3 months, 6 months and 12 months
  six minute walk test (distance reach (m) by walking for 6 minutes)
Change of the Quality of life | pre-pulmonary rehabilitation, 0 months, 3 months, 6 months and 12 months
  COPD assessment test (CAT) (measure the impact of COPD on a person's life, and how this changes over time)
Change in dyspnea | pre-pulmonary rehabilitation, 0 months, 3 months, 6 months and 12 months
  Borg Scale and the medical research center (MRC) scale (scale of 0 to 10 where 0 is no effort and 10 , maximum effort)
Change of Number of hospitalizations | pre-pulmonary rehabilitation, 0 months, 6 months and 12 months
  Self-reported
Change of Number of exacerbations | pre-pulmonary rehabilitation, 0 months, 6 months and 12 months
  We will be able to know to number of exacerbations by the medication taken from the pharmacist of each participant

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633